CLINICAL TRIAL: NCT06254664
Title: Open Label Study to Assess the Effect of Patient Use and Robustness of Tiotropium 18ug Inhalation Powder, Hard Capsule, Zephir Inhaler Device
Brief Title: Open Label Study to Assess the Effect of Patient Use and Robustness of Tiotropium 18ug Inhalation Powder, Hard Capsule,Zephir Inhaler Device
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xiromed LLC (Industry)
Collaborators: Laboratorios Liconsa (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TioDPI PuR-01 (C2A02205)
Record Dates: First submitted 2024-01-30; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Hardness

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tiotropium 18 µg inhalation powder, hard capsule once daily (QD) (Experimental): Interventions:
  Drug: Tiotropium 18 µg inhalation powder, hard capsule
  Device: Zephir inhaler
  Interventions: Drug: Tiotropium 18 µg inhalation powder, hard capsule; Device: Zephir inhaler

INTERVENTIONS:
Drug: Tiotropium 18 µg inhalation powder, hard capsule — Tiotropium 18 µg administered using Zephir inhaler
Device: Zephir inhaler — Tiotropium 18 µg administered using Zephir inhaler

SUMMARY:
An Open Label Study to Assess the Effect of Patient Use and Robustness of Tiotropium 18ug Inhalation Powder, Hard Capsule, Inhaler Device. Zephir inhaler robustness will be assessed by in vitro testing of the Zephir inhaler after 12 weeks of patient use

ELIGIBILITY:
Inclusion Criteria (abbreviated):

1. Capable of understanding the requirements, risks, and benefits of study participation, and as judged by the Investigator, capable of giving written informed consent.
2. Male or non-pregnant female subjects between 40 to 75 years of age at Screening Visit (Visit 1) diagnosed with COPD.
3. General good health (except the COPD diagnosis) and free of any concomitant conditions that would put the subject at increased risk during the study as per the discretion of the Investigator.
4. An established physician diagnosis of COPD as defined by GOLD 2022.
5. At Screening Visit, post-bronchodilator FEV1≤80% and ≥40% of predicted normal values as per Global Lung Function Initiative (GLI-2012) - and post-bronchodilator FEV1/FVC ratio ≤0.70.
6. Current COPD Therapy: Subjects must be on stable regimens of one of the following for at least 8 weeks prior to screening (Visit 1):

   * Long-acting muscarinic antagonist (LAMA)
   * LAMA+LABA
   * Inhaled corticosteroids + LAMA
7. Current or ex-smokers with ≥10 pack-year smoking history (Note: Pack- Year= (cigarettes smoked per day x years smoked)/20)).
8. No occurrence of an upper or lower respiratory tract infection 14 days before Screening Visit.
9. No COPD exacerbation, defined as any worsening of COPD requiring an emergency department visit or hospitalization, or the use of antibiotics (strong CYP450 3A4 inhibitors with ≥ 14 days of acute non-respiratory
10. Ability to adequately use the Test inhaler.

Exclusion Criteria (Abbreviated):

1. Treatment for mild-moderate COPD exacerbations within 4 weeks prior to the Screening Visit (Visit 1) or more exacerbations in the last year.
2. Hospitalization for COPD or pneumonia within 12 weeks prior to the Screening Visit (Visit 1).
3. History of a life-threatening COPD episode that required intubation and/or was associated with hypercapnia, respiratory arrest, hypoxic seizures, or mMRC (Modified Medical Research Council) dyspnea Grade 4.
4. Acute (viral or bacterial) upper or lower respiratory tract infection, sinusitis, rhinitis, pharyngitis, urinary tract infection or illness within 4 weeks prior to the Screening Visit (Visit 1).
5. Subjects with a history of asthma or a clinical diagnosis of asthma, allergic rhinitis, or atopy; a total blood eosinophil count above 600/mm3.
6. Historical or current evidence of a clinically significant disease
7. Have any of the following conditions that, in the judgment of the Investigator, might cause participation in this study to be detrimental to the subject.
8. A subject must not have any clinically significant, uncontrolled condition, or disease state that, in the opinion of the Investigator, would put the safety of the subject at risk through study participation.
9. History of allergy or hypersensitivity to anticholinergic/muscarinic receptor antagonist agents, beta-2 adrenergic agonists, lactose/milk proteins, or specific intolerance to aerosolized tiotropium-containing products or its derivatives.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
In vitro Measurement of Emitted Dose | 3 weeks

CONTACTS AND LOCATIONS:
Locations (9):
- United States (8):
  - Vanguard Clinical Research, LLC, Fort Myers, Florida
  - Clinical Research Solutions - Orlando, Kissimmee, Florida
  - Clintex Research Group, Miami, Florida
  - My Preferred Research LLC, Miami, Florida
  - Research Institute of South Florida, Inc., Miami, Florida
  - Vista Health Research, Miami, Florida
  - Greater Providence Clinical Research, LLC, Cranston, Rhode Island
  - Inquest Clinical Research, LL, Cypress, Texas
- Cliantha Research, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: Undecided